CLINICAL TRIAL: NCT06922396
Title: Predictors of Mortality Among Patients With Head Trauma
Status: Recruiting | Type: Observational
Sponsor: Ayman Mahmoud Alsayes (Other)
Responsible Party: Sponsor-Investigator, Ayman Mahmoud Alsayes, Predictors of Mortality among Patients with Head Trauma, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: Mortality prediction in TBI
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: The Usefulness of Specific Scores in Predicting Mortality of Patients With Head Trauma in ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors group
  Interventions: Other: Parameters on admission
- Non survivors group
  Interventions: Other: Parameters on admission

INTERVENTIONS:
Other: Parameters on admission — A: Parameters on admission:
  * Age.
  * Sex.
  * Comorbidities (DM, HTN, CKD, IHD, Liver Disease)
  * Mode of trauma.
  * Laboratory data (RBS, INR, AST, ALT, Urea, Creatinine, WBC ,HB, CK, Myoglobin).
  * Ct brain findings.
  * Scoring system (GCS, RTS, APACHE II).
  B: Parameters after 2 weeks:
  * Days on Mechanical Ventilation.
  * Medical or surgical management.
  * Complications (Pneumonia, DVT, septic shock, Pulmonary embolism, ARDS).
  Other Names: Parameters after 2 weeks

SUMMARY:
Evaluate the usefulness of the APACHE II (Acute Physiology and Chronic Health Evaluation II), RTS (Revised trauma score), GCS (Glasgow Coma Scale) scores and various variables as age, sex, lab.data and complications in predicting mortality of patients with traumatic brain injury (TBI) in the intensive care unit (ICU).

DETAILED DESCRIPTION:
Head injuries are a major cause of morbidity and mortality through out the world. It is estimated that 69 million people suffer from Traumatic Brain Injury (TBI) from all cases per year .

Current estimates suggest that about 4.48 million people lose their lives due to injuries which accounts for 8% of all deaths globally. Of these, an estimated 2 million deaths were attributed to the TBI, and the burden was concentrated in developing countries due to limited access to advanced life-sustaining measures after trauma .

In low-and middle-income countries, head injury patients have worse outcomes than patients in high-income countries . Several studies in Africa have found that death rates from head injury range from 4.2% to 35% .

Evidence suggests that the possible causes for the high mortality rate could be older age, male gender,low GCS, and cause of injuries are likely non-modifiable risk factors and hypoxia, hypotension, hyperthermia, hypo or hyperglycemia, and did not undergo surgery or poor adherence to management guidelines are possible modifiable risk factors .

Clinical presentation of patients and advanced rescue care by emergency teams are crucial factors to determining favorable outcomes. Accordingly, non-surgical management should emphases on rapid transportation, avoiding hypotension and hypoxia, hyperthermia, and medical management to reduce brain edema .

Accurate determination of the prognosis is crucial for the practitioners, in order to optimize and personalize treatment strategies. There is a degree of uncertainty in clinicians' expectations of patient outcomes, and prognostic models can help improve these expectations by providing probabilities of specific outcomes. Compared with the experience of physicians to judge the prognosis of patients, objective prognostic models would be able to give more accurate projections about specific variables such as number of hospitalizations and deaths .

The predictors of mortality modules used are GCS, APACHE II and RTS scores. GCS provides an objective recording of the state of consciousness of a person, which is the only variable referring to brain function in the APACHE II score. APACHE II score was primarily designed to predict mortality in ICUs. The famous models: the International Mission for Prognosis and Analysis of Clinical Trials (IMPACT) model and the Corticosteroid Randomization After Significant Head Injury (CRASH) model were weighted towards mixed TBI (moderate and severe TBI).

The management of TBI patients should be followed intracranial pressure monitoring is suggested to reduce post-traumatic death in the hospital within two weeks .

Unfortunately, pre hospital care is not well established and hospitals are not well equipped;this can increase the risk of secondary brain injury due to hypotension and hypoxia .

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute traumatic brain injury older than 16 years where presented in emergency department within 24 hours of trauma with a Glasgow coma scale less than 15

Exclusion Criteria:

* o Post cardiac arrest

  * Patients with GCS=3.
  * Patients with associated advanced cervical spine, maxillofacial, severe chest trauma.
  * Patients with previous neurological disorders

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 140 patients admitted to I.C.U during the period of the study, all the studied populations will diagnosed to have an acute traumatic brain injury (TBI).
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
The studied patients will be observed for 1 month and mortality will be recorded. | average 6 to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Medicine , Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No